CLINICAL TRIAL: NCT04833283
Title: The Effects of Intermittent Hypoxic-hyperoxic Preconditioning for Patients Undergoing Cardiac Surgery Using Cardiopulmonary Bypass and Its Impact on Postoperative Complications.
Brief Title: The Effects of Intermittent Hypoxic-hyperoxic Preconditioning for Patients Undergoing Cardiopulmonary Bypass.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 101499310010796
Record Dates: First submitted 2021-03-23; First posted 2021-04-06 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-05

CONDITIONS: Valvular Heart Disease; Aortic Arch Aneurysm; Surgery
Keywords: cardiac pulmonary bypass; reperfusion; interval hypoxic-hyperoxic training; preconditioning; valvular heart disease, aortic arch aneurysm
MeSH Terms: conditions — Heart Valve Diseases; Aneurysm, Aortic Arch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group intermittent hypoxic-hyperoxic training (Experimental): the intervention group is patients performing intermittent hypoxic-hyperoxic training before operation. ReOxy Cardio device, intermittent hypoxic-hyperoxic training ( IHHT)
  Intervention Description: Perform 4 trainings daily of intermittent hypoxic hyperoxic trainings before surgery, using 40 min trainings periods, the patient will receive air with reduced oxygen content (12 %) through a mask under constant monitoring of heart rate (HR) and SpO2. As a safety measure, minimal SpO2 was set at 82 % and maximal accepted increase of heart rate was set to + 50 % of the initial HR. When these values would be reached, the supply of oxygen automatically switched to a hyperoxic gas mixture (35% - 40% O2), inhaling of which would be continued until SpO2 reached 100% (even if SpO2 would be lower before the procedure), which, depending on the rate of saturation reduction, will takes 1 to 3 min (mean 1 min and 50 s).
  Interventions: Device: ReOxy Cardio device, intermittent hypoxic-hyperoxic training ( IHHT)
- the control group (Placebo Comparator): intermittent hypoxic-hyperoxic training control group will be identical to the main group, also underwent four daily procedures before surgery using 40 min training periods with simulation of intermittent hypoxic-hyperoxic trainings by using the same equipment, whereas moistened air will be delivered through a placebo mask
  Interventions: Device: ReOxy Cardio device

INTERVENTIONS:
Device: ReOxy Cardio device, intermittent hypoxic-hyperoxic training ( IHHT) — Perform 4 trainings daily of intermittent hypoxic hyperoxic trainings before surgery, using 40 min trainings periods, the patient will receive air with reduced oxygen content (12 %) through a mask under constant monitoring of heart rate (HR) and SpO2. As a safety measure, minimal SpO2 was set at 82 % and maximal accepted increase of heart rate was set to + 50 % of the initial HR. When these values would be reached, the supply of oxygen automatically switched to a hyperoxic gas mixture (35% - 40% O2), inhaling of which would be continued until SpO2 reached 100% (even if SpO2 would be lower before the procedure), which, depending on the rate of saturation reduction, will takes 1 to 3 min (mean 1 min and 50 s).
  Arms: the intervention group intermittent hypoxic-hyperoxic training
Device: ReOxy Cardio device — Perform 4 trainings daily of intermittent hypoxic-hyperoxic trainings before surgery, using 40 min trainings periods, whereas moistened air will be delivered through a mask under constant monitoring of heart rate (HR) and SpO2.
  Arms: the control group

SUMMARY:
The aim of the study is to evaluate the effects of intermittent

hypoxic-hyperoxic training (IHHT) to protect myocardium against perioperative

myocardial injury during cardiac surgery using cardiopulmonary bypass.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized controlled clinical trial, which will involve patients over 18 years old who would be recruited consecutively during pre-admission consultation at the I.M Sechenov First Moscow State Medical University Cardiac Surgery Department. All patients with a diagnosis of valvular heart disease, or aortic arch disease and indications for cardiac surgery, according to the European Society of Cardiology/European Association for Cardio-Thoracic Surgery guidelines.

Five days before the operation, patients will be randomly assigned into two groups using a computer-generated randomization table: intermittent hypoxic-hyperoxic training and an intermittent hypoxic-hyperoxic training control group. For both groups laboratory testing (specific biomarkers - C-reactive protein, troponin I, fatty acid-binding protein (FABPs) and lactate) will be performed before training and after the surgery, and the hypoxic-inducible factor (HIF 1 alpha) would be implemented before and after the trainings.

Patients in the intermittent hypoxic-hyperoxic training group will undergo four daily procedures of interval hypoxic-hyperoxic training before cardiac surgery, using a normobaric device to obtain hypoxic and hyperoxic gas mixtures (ReOxy Cardio; Aimediq S.A., Luxemburg, Registration certificate in RU P3H 2014/1486). Before the start of the training, each patient would undergo a hypoxic test to assess the individual response to hypoxia, and to determine the rate of reduction of blood oxygen saturation (SpO2) with a finger pulse oximeter (Masimo SET, measurement accuracy ±2%). During 5 minutes the patient will receive air with reduced oxygen content (12%), through a mask under constant monitoring of the heart rate (HR) and SpO2. As a safety measure, minimal SpO2 would be set at 82% and maximal accepted increase of heart rate would be set to +50% of the initial heart rate. When these values would be reached, the supply of oxygen automatically would be switched to a hyperoxic gas mixture (35%-40% O2), inhaling of which would be continued until SpO2 reached 100% (even if SpO2 was lower before the procedure), therefore depending on the rate of saturation reduction, will be taken 1 to 3 minutes (mean 1 min and 50 seconds). The intention is to create hyperoxic arterial oxygen tension and not to simply reduce the time required to recover from hypoxia. Intermittent hypoxic hyperoxic training would be considered successful if there were no significant side effects during the procedure such as angina pain, loss of consciousness, severe dizziness or other variants of significant subjective deterioration of the patient's condition. In the case of successfully passing the test, patients will proceed to the basic intermittent hypoxic hyperemic training. During the training, the hypoxic gas mixture will be given to the patient again in intermittent mode, based on the individual test parameters and alternating with the supply of a hyperoxic gas mixture. One cycle of the procedure consists of hypoxic and hyperoxygenated intervals, the duration of which will be regulated automatically according to the biofeedback principle, based on monitoring of individual values of SpO2 and heart rate. The duration of the hypoxic period ranges from 3 to 5 minutes, and the duration of the hyperoxic period ranges from 1 to 3 minutes, depending on the SpO2 recovery rate. The total time of the hypoxic gas mixture inhaled during one procedure will be 20-30 min. A final training would be conducted in the evening before the surgery. Patients in the intermittent hypoxic-hyperoxic training - control group also will undergo four daily procedures before surgery, using 40 min training periods with simulation of intermittent hypoxic-hyperoxic training by using the same equipment, the patient receives moistened air through a placebo mask under constant monitoring of heart rate and SpO2. Only the person who will conduct the training would know about the patient's allocation to a particular intervention group, the anesthesiologists and cardiac surgeons will not have access to this information. Episodes of cardiac arrhythmias, hypotension with a need for inotropic drug prescription, changes in electrocardiogram, pulse values and blood pressure levels will be recorded during surgery and the postoperative period.

Patients will be monitored for 7 days in the hospital, and 30 days after discharge to evaluate the complications.

Differences between groups will be assessed using the unpaired Student's t-test or the one-tailed Anova test followed by the Bonferroni post-test. Baseline corrected logistic regression models will be used to estimate the training effect in relation to primary and secondary endpoints. Statistical significance will be set at 0.05 to test hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written consent to participate in the study 2. Male or female patients over 18 years 3. Indications for planned replacement of the aortic or mitral valves or operations on the aortic arch.

Exclusion Criteria:

* 1. Individual intolerance to the intermittent hypoxic-hyperoxic training

  2. Acute coronary syndrome after hospitalization and before the surgery

  3. The presence of an acute infectious process after hospitalization and before the surgery (fever, leukocytosis with a shift leukocyte formula to the left, increased erythrocyte sedimentation rate (ESR), increased C-reactive protein)

  4. Uncompensated hypertension at the time of the procedure (systolic blood pres-sure more than 160 mm Hg, diastolic blood pressure more than 110 mm Hg)

  5. Loss of consciousness, severe dizziness

Non-inclusion criteria:

1. Occlusive atherosclerotic disease of lower limbs,
2. Acute coronary syndrome within 4 weeks before entry
3. Preoperative renal insufficiency (serum creatinine higher than 200 mmol/L),
4. Acute infectious diseases
5. Partial and secondary generalized forms of epilepsy,
6. Uncompensated hypertension (Blood pressure at the time of the procedure: systolic blood pressure more than 160 mm Hg, diastolic blood pressure more than 110 mm Hg)
7. Severe bronchial asthma with the development of respiratory failure of the II-III degree and individual intolerance to oxygen deficiency.

9. Severe hepatic impairment (class C child-Pugh) Intervention type

10. Mental illness (if patients are not capable of understanding the nature, significance and implications of the clinical trial)

11. Myocardial insufficiency as a component of multiple organ failure in decompensation of liver and kidney diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Death from a cardiac cause | The first 30 days from the date of discharge
  Death from cardiac causes during the current hospitalization or 30 days after discharge
Myocardial infarction | through study completion, an average of 1 month after discharge
  Myocardial infarction after current surgery and one month after discharge
Stroke | through study completion, an average of 1 month after discharge
  Stroke in postoperative period until the date of the discharge

SECONDARY OUTCOMES:
Electrocardiogram deterioration caused by myocardial ischemia; | through study completion, an average of 1 month after discharge
  Electrocardiogram deterioration caused by myocardial ischemia (ST segment elevation or depression, Q wave, negative T wave ) during hospitalization or 30 days after discharge
Angina pectoris - typical chest pain III - IV functional class (Canadian Cardiovascular Society classification) | through study completion, an average of 1 month after discharge
  Having an angina pectoris during hospitalization or 30 days after discharge
Documented episodes of atrial fibrillation/ atrial flutter. | through study completion, an average of 1 month after discharge
  Documented episodes of atrial fibrillation or atrial flutter during hospitalization or 30 days after discharge
Ventricular proarrhythmia requiring additional therapy | through study completion, an average of 1 month after discharge
  Detection of ventricular proarrhythmia during hospitalization or 30 days after discharge
Atrioventricular block 2-3 degrees | through study completion, an average of 1 month after discharge
  Atrioventricular block 2-3 degree during hospitalization or 30 days after discharge
Episodes of hypotension requiring additional therapy | through study completion, an average of 1 month after discharge
  Episodes of hypotension (systolic blood pressure of less than 90 mmHg/ diastolic of less than 60 mmHg) requiring additional therapy during hospitalization or 30 days after discharge
Length of stay in the intensive care unit | through study completion, an average of 1month

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Hospital №1, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Data disclosure is not permitted by the local ethics committee. For more information about the study, you need to contact the principal investigator.